CLINICAL TRIAL: NCT04170881
Title: Daycare Environmental Exposure to Cleaning Products and Respiratory Health in Young Children and Daycare Workers
Brief Title: CRESPI - Respiratory Health of Children in Daycare
Acronym: CRESPI
Status: Active, not recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Centre Scientifique et Technique du Bâtiment (Unknown); EPICONCEPT (Unknown); Ecole des Hautes Etudes en Santé Publique (Other); ANSES (Other); ADEME (Unknown); National Research Agency, France (Other); Agence Regionale de Sante d'Ile de France (Other Government); Fondation de France (Other)
Responsible Party: Sponsor
Other Study IDs: C 18-05
Record Dates: First submitted 2019-11-05; First posted 2019-11-20 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Respiratory Health
Keywords: cleaning products; respiratory health; young children; nursery workers; nursery environment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CHILDREN: Children from involved daycares (Paris region)
  Interventions: Other: Exposed/non exposed - Epidemiology
- WORKERS: workers in involved daycares (Paris region)
  Interventions: Other: Exposed/non exposed - Epidemiology

INTERVENTIONS:
Other: Exposed/non exposed - Epidemiology — visit of daycares and environmental measurement will be performed

SUMMARY:
CRESPI - RESPIratory health of Children in daycare

The CRESPI study, will be a cohort of 1500/2000 children attending daycare in Paris region, and will be initiated in November 2019.

The aim of the project is to study the impact of environmental exposures to cleaning products and disinfectants on respiratory health of infants and toddlers (< 3 years) in daycares

Two specific aims were defined:

1. evaluate environmental exposure to cleaning products by complementary and innovative tools: air quality measurements in daycares, specific standardized questionnaire, identification of compounds of the products via a database and a Smartphone application to scan bar codes and inform on product use
2. evaluate the impact of early exposure in daycares and at home on respiratory health of young children

DETAILED DESCRIPTION:
Context

Exposure to cleaning products is an emergent risk factor for respiratory health of children. In some studies, an association has been observed between the use of these products in households and wheezing in young children (<18 months). However, the specific chemical substances associated with health hazards remain poorly known. A few studies suggested associations between some specific organic volatile compounds (aldehydes, aromatics) and asthma but only one study has been conducted in young children (<3 years). Detergents/disinfectants may contain sensitizers, irritants and endocrine disrupters. Children who attend daycares may be particularly exposed: cleaning tasks are often performed in their presence; moreover, babies and young children often put objects (eg, toys) in their mouths and might be exposed through various routes (ingestion, inhalation, skin). The importance of studying the health impact of early life environmental exposures has been emphasized, especially in the context of the Developmental Origins of Health and Diseases (DOHaD) research. However, few studies have focussed on environmental exposures in nurseries in relation to children's respiratory health.

The originality of the CRESPI cohort lies in the fact that no epidemiological survey focussed on: 1) the effect of early exposure to cleaning products in daycares on respiratory health in first years of life; 2) the use of complementary and innovative tools to improve evaluation of such exposures, via a Smartphone application and measurements of pertinent volatile (VOCs) and semi-volatile (SVOCs) organic compounds. 3) the use of complementary and innovative tools to improve evaluation of children respiratory health, via a Smartphone application

Methods

The project CRESPI (http://crespi.vjf.inserm.fr/) is to set up an epidemiological survey among young children attending daycares. A sample of 400 daycares (30-40 children/daycare) in Ile-de-France (Paris region) has been drawn from a national file. We hypothesise that the acceptance rate of daycares will be of 25% and those of parents at least of 50% (see French OQAI study 2011), with an expected population of 1500 to 2500 children.

Each daycare will be visited by trained interviewers to : i) precise the objectives of the study to the parents/workers in the daycare and give all material to collect data (questionnaire, smartphone); ii) collect dust samples (to measure SVOCs; triclosan, muscs ...) via an adapted vacuum cleaner and install measuring equipment to evaluate air quality (VOCs; ammoniac, glycol ethers ...); iii) collect information on the building (surface, ventilation …) and activities of workers including a calendar of cleaning tasks in rooms (toilets, bedroom ...) and surface (toys, windows, toddler beds …).

A standardized questionnaire (http://crespi.vjf.inserm.fr/), as previously used in a parent-child cohort (sepages.inserm.fr), collecting information on the use of products, respiratory health and potential confounders will be completed by the parents. Respiratory health of the children will also be evaluated by a group of experts (paediatricians) using information available from medical records (children's health booklets).

This project will take full advantage of innovative tools, i.e. Smartphone applications, to evaluate 1) exposures : workers and parents will scan bar-codes of products used, in the nursery and at home, and respond to a short questionnaire about their use, and 2) respiratory health of children, with monthly follow-up.

Statistical analyses of the data will evaluate the associations between exposures and respiratory health of children, after adjustment for potential confounders.

ELIGIBILITY:
Inclusion Criteria:

Children :

* aged from 2 months to 3 years (< 4 years) attending daycares in Paris region, among those which accepted to participate to the CRESPI study
* signed and dated written informed consent form obtained from at least one parent

Nursery workers :

* all those who accepted to participate
* signed and dated written informed consent form obtained

Exclusion Criteria:

Children and workers : if it is impossible for them (parents or workers) to understand French langage and/or to follow the questionnaire of the study

Children

* both parents less than 18 years old
* parents subjected to a legal protection measure or deprived of liberty by judicial or administrative decision
* if at least two children of the same familly attended the same daycare, only the youngest one will be included. In case of twins or triplets, only one children will be chosen at random.

Ages: 2 Months to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: CRESPI is an epidemiological survey among young children - aged from 3 months to 3 years old - attending daycares and daycare workers. A random sample, drawn from a national file, of 400 nurseries in Paris region have been selected. Out of them, the 100 first daycares (30-40 children/nursery) who accepted to participated will be visit.
  The CRESPI project will include detailed characterization of chemical exposures in 100 daycare centers evaluated during a one-day visit, between 2019 and 2021. We expected to enrol around 1500/2000 children and 600/800 adults workers (18-65 years old).
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-12-03 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2029-12-03 (Estimated)

PRIMARY OUTCOMES:
Current wheezing | at inclusion (2019-2021)
  'Current wheezing' phenotypes will be defined by questionnaires (paper, smartphone, web), based on responses to epidemiological standardized questionnaires and in accordance with definitions used in international studies:
  * wheezing in the last 12 months
  * severe wheezing in the last 12 months (defined by wheezing in the last 12 months with use of inhaled corticosteroid and/or the need for hospital-based care [emergency department visit and/or hospitalization due to bronchiolitis wheezy bronchitis or asthma attacks] in the last 12 months)
  * recurrent wheezing (at least 3 wheezing episodes in the last 12 months).
Longitudinal wheezing | at inclusion (2019-2021), every month by a smartphone application (during 1 year after inclusion), every 6 months by questionnaires (2021 to 2023)
  Longitudinal wheezing phenotypes will be defined by longitudinal latent class analysis (statistical clustering approach), making full use of data collected by questionnaire during follow-up (first monthly and then every six months), from infancy to age 4-years.

SECONDARY OUTCOMES:
Current cough | at inclusion (2019-2021)
  Cough in the last 12 months defined by a standardised questionnaire will also be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Le Moual, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France; Orianne Dumas, PhD, Study Chair — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Nicole LE MOUAL, Villejuif, France

IPD SHARING:
Plan to Share IPD: No